CLINICAL TRIAL: NCT03426670
Title: HIV Self-Testing to Empower Prevention Choices in Sex Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: University of Washington (Other); Massachusetts General Hospital (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ST/189/2017
Record Dates: First submitted 2018-01-10; First posted 2018-02-08 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: HIV/AIDS
Keywords: HIV self-testing; Pre-exposure prophylaxis; Sex workers
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Randomization in a 1:1 ratio to either monthly HIVST with quarterly in-clinic testing (intervention) or quarterly in-clinic HIV testing (standard of care).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OraQuick HIV Self-Test (Active Comparator): Sex workers in the intervention arm will be instructed to self-test before starting each monthly course of PrEP. HIV Self-testing will be performed during the months between scheduled quarterly visits.
  Interventions: Device: OraQuick HIV Self-Test
- In-clinic testing (No Intervention): All study participants will receive quarterly in-clinic HIV testing as standard-of-care.

INTERVENTIONS:
Device: OraQuick HIV Self-Test — OraQuick® HIV Self-Test is an in-vitro diagnostic medical device that is used for self-testing of antibodies for HIV-1 and HIV-2 in oral fluid. This test is intended as an aid to detect antibodies to HIV-1 and HIV-2 from infected individuals.
  Arms: OraQuick HIV Self-Test

SUMMARY:
Transgender, male, and female sex workers are 49, 21 and 14 times as likely to be HIV-infected as other adults in the general population. In Uganda, sex workers have high HIV seroprevalence (35-37%) and account for 10% of new HIV infections. Two robust, evidence-based, self-controlled HIV prevention tools are available -- HIV self-testing (HIVST) and antiretroviral pre-exposure prophylaxis (PrEP) -- but these are not currently well utilized among sex workers. HIVST and PrEP are complementary tools that could be combined to build self-efficacy and empowerment, increase PrEP adherence and reduce sexual risk behaviors. However, research is needed to show how combination HIVST and PrEP may have a synergistic impact on uptake and use of each prevention intervention. The investigators will conduct a randomized trial among sex workers initiating PrEP in Uganda to test if HIV self-testing increases PrEP adherence among HIV-uninfected sex workers (Aim 1), changes sexual risk behavior in sex workers taking PrEP (Aim 2), and influences prevention choices among sex workers and their partners (Aim 3). The investigators will use novel technologies (real-time electronic monitoring with Wise pill technology and mobile phone surveys) to characterize patterns of PrEP adherence, and assess how use of HIVST and PrEP aligns with sexual risk behaviors. Additionally, the investigators will conduct in-depth qualitative interviews to explore the mechanisms through which combined HIVST and PrEP delivery may be synergistic and empowering. This study will be the first to jointly evaluate HIVST and PrEP in sex workers.

DETAILED DESCRIPTION:
This is a randomized clinical trial of HIV-uninfected transgender, female, and male sex workers. The overall goal is to test if HIV self-testing increases PrEP adherence (Aim 1), changes sexual risk behavior (Aim 2), and influences HIV prevention choices (Aim 3) in HIV-uninfected sex workers and their partners. For Aim 1, the investigators will recruit HIV-uninfected sex workers in Kampala, Uganda and randomize them to the intervention (monthly HIVST with quarterly clinic-based testing) or the control arm (quarterly clinic-based testing). Study participants will be trained how to use and interpret HIVST and be provided with 4 kits at enrollment and each quarterly visit: 2 kits for own use and 2 for sexual partners, with additional kits provided as needed. They will be instructed to self-test before opening a new PrEP bottle. The investigators will use Wise pill technology to evaluate patterns of PrEP use, and mobile phone interviews to assess HIVST use and confidence in PrEP effectiveness. The investigators will conduct Aim 2 within the randomized trial in Aim 1 and test whether HIVST changes sexual risk behavior. The investigators will use mobile phone interviews and semi-structured questionnaires to collect the behavioral data. In Aim 3 the investigators will use qualitative methods to assess how HIVST empowers use of HIV prevention interventions among sex workers and their partners.

Aim 1: To test if HIV self-testing versus clinic-based testing increases PrEP adherence among HIV-uninfected sex workers.

Approach: To evaluate the impact of HIVST on PrEP adherence, the investigators will randomize 110 HIV-uninfected transgender, female and male sex workers initiating PrEP in a 1:1 ratio to either monthly HIVST with quarterly in-clinic testing (intervention) or quarterly in-clinic HIV testing (standard of care). PrEP medications will be dispensed quarterly. Sex workers in the intervention arm will be instructed to self-test before starting each monthly course of PrEP. In this study, participants will receive counseling on the importance of strict PrEP adherence for HIV protection.

Hypothesis: Monthly HIVST will empower HIV prevention and motivate PrEP adherence among HIV-uninfected sex workers.

Aim 2: To test the effect of HIV self-testing on sexual risk behavior in sex workers taking PrEP.

Approach: Within the randomized trial in Aim 1, the investigators will provide HIVST kits to sex workers for own use, and with partners (primary and commercial). The investigators will use monthly live phone interviews and semi-structured questionnaires to collect data on high-risk sexual behaviors (e.g. sexual frequency, unprotected sex).

Hypothesis: Use of HIVST will be associated with decreased frequency of unprotected sex and sexually transmitted infections.

Aim 3: To explore how HIV self-testing influences prevention choices among sex workers and partners.

Approach: The investigators will conduct in-depth interviews with sex workers and their primary and commercial partners to assess perceptions and experiences with HIVST, explore how HIVST influences status disclosure, behavior change and PrEP use, and to better understand how mobile technology can be leveraged to motivate repeat testing in individuals at high ongoing risk of HIV.

Hypothesis: HIVST will empower sex workers to adopt protective behaviors, facilitate partner testing, and efficiently identify individuals with undiagnosed HIV infection.

ELIGIBILITY:
Inclusion Criteria:

* Exchanged sex for goods or money at least once in the prior month
* Able and willing to provide written informed consent
* HIV-uninfected based on negative HIV rapid tests according to the national Uganda algorithm
* Adequate renal function (normal creatinine levels; calculated creatinine clearance ≥ 60ml/min)
* Not infected with Hepatitis B virus (negative HBsAg test)
* Not enrolled in HIV prevention trial currently or within the past year
* Not currently using PrEP
* Willing to remain in the study for the next 12 months
* Own a mobile phone for personal use
* Have regular access to electricity for charging a mobile phone

Exclusion Criteria:

* A physical or mental condition that prohibits informed consent and/or participation in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender
Enrollment: 110 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
PrEP adherence as measured by Wisepill electronic adherence monitors and intra-cellular tenofovir drug levels | 12 months
  Comparison of adherence outcomes by randomization arm

SECONDARY OUTCOMES:
High-risk sexual behaviors as measured by frequency of unprotected sex and sexually transmitted infections | 12 months
  Comparison of self-reported unprotected sex and sexually transmitted infections by randomization arm
Proportion of sex workers using self-test kits | 12 months
  Proportion of sex workers randomized to HIV self-testing using HIV self test kits
Diagnostic accuracy of HIVST in oral PrEP users | 12 months
  Proportion of false negative HIV self-test tests
Self-reported confidence in PrEP effectiveness as measured by monthly questionnaires | 12 months
  Proportion who believe PrEP is effective in preventing HIV infection

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Mujugira, MBChB, PhD, Principal Investigator — Center Head
Locations (1):
- Infectious Diseases Institute,Makerere University College of Health Sciences, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No